CLINICAL TRIAL: NCT06755658
Title: RDW (red Cell Distribution Width) and What Has Happened to the Platelets. is There an Association of RDW and Platelet Kinetics (PLTs and MPV/PLT Ratio), with Survival Outcome in Covid -19 Hospitalised Patients?
Brief Title: RDW, Platelet Kinetics and Survival Outcome in Covid-19 Hospitalized Patients.
Acronym: HEMLABFORCOV19
Status: Active, not recruiting | Type: Observational
Sponsor: Sismanoglio General Hospital (Other)
Responsible Party: Principal Investigator, DESPOINA GEORGIADOU, MD, HEMATOLOGIST, Sismanoglio General Hospital
Other Study IDs: 16526/23-08-2023
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Infection by SARS-COV-2
Keywords: COVID-19; SARS-COV-2; RDW; PLTs; MPV/PLT ratio; Survival; Coagulation
MeSH Terms: conditions — COVID-19; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- A Cohort of patients with COVID-19 hospitlaized: Study admission criteria
  1. Adults over 18 years old, who required hospital treatment for more than 24 hours for SARS-COV -2 infection, confirmed by molecular testing (rRT - PCR) and within one (1) month of the positive test for covid-19 diagnosis.
  2. Patients directly admitted to the General Hospital Sismanoglio - A.Fleming or coming for admission and continuance of treatment for covid-19 disease, from other hospitals of 1st Health Region of Attica, where diagnosed with covid-19 disease first, with clinical information notes and laboratory data at their admission and hospitalization.
  3. Patients without myelodysplastic syndrome, iron deficiency or low values of B12, folic acid.

SUMMARY:
This is a retrospective, non-interventional nor experimental study conducted at the General Hospital of Athens "Sismanoglio - A. Fleming / A. Fleming Hospital Unit" in hospitalized covid-19 patients who will be tested for RDW, PLT and MPV / PLT ratio, parameters in routine complete blood counts, in relation to mortality risk, during the years 2020-2021, since November 2020, when the hospital was designated, by Ministerial decision, exclusively for the treatment of covid-19 patients until June 2021, a period corresponding to the prevalence of the delta subtype, according to the local epidemiological surveillance of the National Public Health Organization of Greece. (https://eody.gov.gr/).

DETAILED DESCRIPTION:
INTRODUCTION -CONCEPTION OF THE IDEA OF THE STYDY The erythrocytic index RDW is a parameter of red blood cells, expresses anisocytosis in the red blood population (11.5-14.5%) and its values are determined in the routine blood count of 25 parameters. (1,2,3)The medical literature shows that a raised RDW is associated with an increased risk of death in a number of pathological conditions, heart disease, lung disease, stroke, sepsis, cancer.(4,5,6,7) With the burst of publications concerning Covid-19 disease, there is extensive reference to the relationship of RDW with the severity and mortality of the disease. (8,9,10,11,12,13) Similarly, lower platelet counts (PLTs) - thrombocytopenia are common in Covid-19 disease, through a variety of mechanisms and are related to its severity and outcome, as reported in a systematic review of 24 studies,(14) but also in a meta-analysis of 9 studies where, despite the great heterogeneity among them, the more sizeable drop of platelets was observed in non-survivors.(15,16,17) In addition, although covid-19 disease affects mainly the respiratory system and can lead to respiratory failure, it also comes with a high number of thromboses with raised D-dimers and findings of micro thrombosis in the lungs or other organs of the affected deceased. To the coagulopathy of covid-19 disease that resembles but is not identical to other coagulation disorders such as sepsis-DIC (SIC/DIC), hemophagocytic syndrome (HPS), antiphospholipid syndrome (APS) and thrombotic microangiopathy (TMA),(18) contributes, the overactivation of platelets and immunothrombosis that often occurs in severe covid-19 disease.(19) In the systematic review by Daniels and colleagues, 32 studies were found that examined markers related to platelet size (Platelet Volume Indexes, PVI) in relation to the severity or mortality of covid-19 disease.(20) The PVI parameters in these studies included, in addition to platelet count PLT and MPV, others, such as PDW, P-LCR, LMR, MPR, to a varying degree and combination. The results showed a general trend that high values of these markers are associated with disease severity and mortality.(20) The 14 studies of the review, reported significant differences in baseline PVI values between severe and mild covid-19 disease, although the longitudinal studies showed varying trends in these platelet markers.(20) In recent years, researchers have been interested in the platelet index MPV/PLT ratio (derived from the ratio of mean platelet volume to platelet count) as a specific marker of platelet-based systemic thrombogenicity.(21,22,23)

AIM OF THE STUDY Our study will examine the relationship of the red cell index RDW, platelet count PLTs and platelet index MPV/PLT ratio, with the risk of mortality in hospitalized patients with SARS-COV2, at entry, discharge, 1st week , 2nd week, as well as the total duration of hospitalization. There are no other reports on this issue in Greece.

If there is a connection and we determine the cut off values we could suggest that Hematology Laboratory may have the potential to assist in early screening and prognosis of COVID-19 disease.

Study Protocol and Patients Group The registered diagnosed with SARS-Cov-2 patients are either directly admitted to the General Hospital Sismanoglio - A.Fleming or coming for continuance of treatment from other hospitals of 1st Health Region of Attica mainly, such as: G.Gennimatas GH, Evangelismos GH, Konstantopoulio GH, Laiko GH, Erythros GH, Alexandra GH, Ippokrateio GH, Attikon GH, with information notes and laboratory data at their admission and hospitalization.

Hematological laboratory testing has been performed on Hematology Analyzers who are subject to Internal and External Quality Control. Regarding the General Hospital Sismanoglio - A. Fleming , the Hematology and Hemostasis Analyzers used, were ADVIA 2-120 , Sysmex Ca-1500, BCS XP by Siemens Healthineers and SYSMEX XE 2100 by Roche Diagnostics.

Patients will be enrolled according to age, gender, comorbidities, covid-19 disease severity, outcome (improvement or death), RDW, PLT, MPV/PLT ratio, parameters, at entry, discharge and mean values of hospitalization duration. To monitor the parameters' trend, the mean values of PLT, MPV/PLT ratio of the 1st and 2nd week of hospitalization will be determined and recorded, the nadir values of PLT, mean and nadir values of lymphocytes (absolute number, percentage% and when), mean and zenith values of CRP and D-dimers, as well as the score for DIC of the deceased, based on ISTH criteria.(24) (Table 1) MPV/PLT ratio is defined and calculated as : : MPV value (fl)x100/ PLT per 1000/μl

The 1st and 2nd week intervals were of interest because between the 7th and 14th day from the onset of the disease, there is a surge of clinical manifestations, with a pronounced increase in inflammatory mediators and cytokines. (25) The values of D-dimer (fibrin degradation products) will be determined and recorded as indicative of endovascular thrombosis and as an independent predictor of mortality risk in covid-19 disease. (26) Lymphocyte values (mean, absolute number, percentage % nadir and when) are also recorded, as lymphopenia is a predominant finding in most severe cases of covid-19 disease (15, 27, 28, 29) and the sequential assessment of lymphocyte dynamics can be predictive of the patient's outcome.(28) The CRP value (mean, zenith and when) is determined and recorded as an indicator of inflammation, especially high in the cytokine storm that can occur in covid-19 patients and is associated with disease mortality. (30) The classification of patients into mild/moderate and severe/critical covid-19 disease was based on the criteria of National Public Health Organization of Greece (EODY).(31) The statistical analysis will be performed by SAS Software for Windows version 9.4 (SAS Institute Inc, NC, USA). For the analysis of variables expressed as numeral values, i.e. quantitative data (e.g., age, RDW, PLTs etc.) and specifically to identify for differences between survivors and non survivors, the statistical analysis is expected to be performed via the Mann-Whitney U test method. However, in case that data do follow the normal distribution as evaluated by the Kolmogorov-Smirnov test then the t-test method will be applied. For the evaluation of differences in the expression of RDW and PLTs and MPV/PLT ratio or other numerical data in various groups (such as different age groups ) the Kruskal Wallis method will be applied and in case of normality will be applied the ANOVA test. Categorical data differences in the study groups (e.g. gender, age groups etc.) will be tested by the x2 test and if required via the Fisher exact test.

The level of statistical significance is set to <0.05 (P <0.05) and all tests will be two-sided.

Finally, the statistical analysis is composed of descriptive statistics, i.e. for numerical variables measures of central values and dispersion such as mean value, median, standard deviation and quartile 1 and 3 (Q1 and Q3) and for categorical variables includes percentages and 95% confidence intervals. For the inferential statistics it will be evaluated the hypothesis that RDW and PLTs, MPV/PLT ratio, values as prognostic markers for the final outcomes of COVID-19 hospitalized patients.

References

1. Dacie and Lewis Practical Haematology 12th Edition - August 11, 2016 Barbara Bain, Imelda Bates, Mike Laffan Red cell indices,Variations in red cell volumes:Red cell distribution width,35-37
2. Naveen Kakkar, Manisha Makkar, Red Cell Cytograms Generated by an ADVIA 120 Automated Hematology Analyzer: Characteristic Patterns in Common Hematological Conditions, Laboratory Medicine, Volume 40, Issue 9, September 2009, Pages 549-555, https://doi.org/10.1309/LM23R7FULSTUJSJD
3. Red Cell Distribution Width (RDW) Test, Medscape Updated: Jun 13, 2022 Choladda Vejabhuti Curry, MD; Chief Editor: Daniela Hermelin, MD
4. Perlstein TS, Weuve J, Pfeffer MA, Beckman JA. Red blood cell distribution width and mortality risk in a community-based prospective cohort. Arch Intern Med. 2009;169(6):588-594. doi: 10.1001/archinternmed. 2009.55 [PMC free article] [PubMed]
5. Bazick HS, Chang D, Mahadevappa K, Gibbons FK, Christopher KB. Red cell distribution width and all-cause mortality in critically ill patients. Crit Care Med. 2011 Aug;39(8):1913-21. doi: 10.1097/ CCM. 0b013e31821b85c6. PMID: 21532476; PMCID: PMC4427349.
6. Patel KV, Ferrucci L, Ershler WB, Longo DL, Guralnik JM. Red blood cell distribution width and the risk of death in middle-aged and older adults. Arch Intern Med. 2009;169(5):515-523. doi: 10.1001/archinternmed.2009.11
7. Zhang L, Yu CH, Guo KP, Huang CZ, Mo LY. Prognostic role of red blood cell distribution width in patients with sepsis: a systematic review and meta-analysis. BMC Immunol. 2020 Jul 6;21(1):40. doi: 10.1186/s12865-020-00369-6. PMID: 32631218; PMCID: PMC7339553.
8. Foy BH, Carlson JCT, Reinertsen E, Padros I Valls R, Pallares Lopez R, Palanques-Tost E, Mow C, Westover MB, Aguirre AD, Higgins JM. Association of Red Blood Cell Distribution Width With Mortality Risk in Hospitalized Adults With SARS-CoV-2 Infection. JAMA Netw Open. 2020 Sep 1;3(9):e2022058. doi: 10.1001/jamanetworkopen.2020.22058. PMID: 32965501; PMCID: PMC7512057
9. Henry BM, Benoit JL, Benoit S, Pulvino C, Berger BA, Olivera MHS, Crutchfield CA, Lippi G. Red Blood Cell Distribution Width (RDW) Predicts COVID-19 Severity: A Prospective, Observational Study from the Cincinnati SARS-CoV-2 Emergency Department Cohort. Diagnostics (Basel). 2020 Aug 21;10(9):618. doi: 10.3390/diagnostics10090618. PMID: 32825629; PMCID: PMC7554711.
10. Lippi G, Henry BM, Sanchis-Gomar F. Red Blood Cell Distribution Is a Significant Predictor of Severe Illness in Coronavirus Disease 2019. Acta Haematol. 2021;144(4):360-364. doi: 10.1159/000510914. Epub 2020 Aug 25. PMID: 32841949; PMCID: PMC7490490.
11. Karampitsakos T, Akinosoglou K, Papaioannou O, Panou V, Koromilias A, Bakakos P, Loukides S, Bouros D, Gogos C, Tzouvelekis A. Increased Red Cell Distribution Width Is Associated With Disease Severity in Hospitalized Adults With SARS-CoV-2 Infection: An Observational Multicentric Study. Front Med (Lausanne). 2020 Dec 11;7:616292. doi: 10.3389/fmed.2020.616292. PMID: 33363191; PMCID: PMC7759673.
12. Lagadinou M, Gkentzi D, Marangos MN, Paliogianni F, Solomou EE. Red Blood Cell Distribution Width: Another Prognostic Factor for COVID-19? Clin Hematol Int. 2021 Apr 10;3(2):69-71. doi: 10.2991/chi.k.210404.001. PMID: 34595468; PMCID: PMC8432399.
13. Banon T, Wortsman J, Ben Moshe S, Gazit S, Peretz A, Ben Tov A, Chodick G, Perez G, Patalon T. Evaluating red blood cell distribution width from community blood tests as a predictor of hospitalization and mortality in adults with SARS-CoV-2: a cohort study. Ann Med. 2021 Dec;53(1):1410-1418. doi: 10.1080/07853890.2021.1968484. PMID: 34409900; PMCID: PMC8381942.
14. Zong X, Gu Y, Yu H, Li Z, Wang Y. Thrombocytopenia Is Associated with COVID-19 Severity and Outcome: An Updated Meta-Analysis of 5637 Patients with Multiple Outcomes. Lab Med. 2021 Jan 4;52(1):10-15. doi: 10.1093/labmed/lmaa067. PMID: 32929506; PMCID: PMC7543465
15. Terpos E, Ntanasis-Stathopoulos I, Elalamy I, Kastritis E, Sergentanis TN, Politou M, Psaltopoulou T, Gerotziafas G, Dimopoulos MA. Hematological findings and complications of COVID-19. Am J Hematol. 2020 Jul;95(7):834-847. doi: 10.1002/ajh.25829. Epub 2020 May 23. PMID: 32282949; PMCID: PMC7262337.
16. Lippi G, Plebani M, Henry BM. Thrombocytopenia is associated with severe coronavirus disease 2019 (COVID-19) infections: A meta-analysis. Clin Chim Acta. 2020 Jul;506:145-148. doi: 10.1016/j.cca.2020.03.022. Epub 2020 Mar 13. PMID: 32178975; PMCID: PMC7102663.
17. Clinical Characteristics of Coronavirus Disease 2019 in China: Guan W, Ni Z, Hu Y, et al. N Engl J Med. 2020 Feb 28 [Online ahead of print] DOI: 10.1056/NEJMoa2002032. J Emerg Med. 2020 Apr;58(4):711-2. doi: 10.1016/j.jemermed.2020.04.004. Epub 2020 Jun 3. PMCID: PMC7266766
18. Iba T, Levy JH, Connors JM, Warkentin TE, Thachil J, Levi M. The unique characteristics of COVID-19 coagulopathy. Critical Care [Internet]. 2020 Jun 18;24. Available from: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7301352/
19. Du F, Liu B, Zhang S. COVID-19: the role of excessive cytokine release and potential ACE2 down-regulation in promoting hypercoagulable state associated with severe illness. Journal of Thrombosis and Thrombolysis. 2020 Jul 16;51(2):313-29.
20. Daniels S, Wei H, van Tongeren M, Denning DW. Are platelet volume indices of clinical use in COVID-19? A systematic review. Front Cardiovasc Med. 2022 Oct 18;9:1031092. doi: 10.3389/fcvm.2022.1031092. PMID: 36329999; PMCID: PMC9623063.
21. Azab B, Torbey E, Singh J, Akerman M, Khoueiry G, McGinn JT, Widmann WD, Lafferty J. Mean platelet volume/platelet count ratio as a predictor of long-term mortality after non-ST-elevation myocardial infarction. Platelets. 2011;22(8):557-66. doi: 10.3109/09537104.2011.584086. Epub 2011 Jun 30. PMID: 21714700.
22. D.H. Shin, S.Y. Rhee, H.J. Jeon, J.Y. Park, S.W. Kang, J. Oh An increase in mean platelet volume/platelet count ratio is associated with vascular access failure in hemodialysis patients PLoS One, 12 (2017), p. e0170357
23. G.H. Oh, S.P. Chung, Y.S. Park, J.H. Hong, H.S. Lee, H.S. Chung, et al. Mean platelet volume to platelet count ratio as a promising predictor of early mortality in severe sepsis Shock, 47 (2017), pp. 323-330
24. Levi M, Toh CH, Thachil J, Watson HG. Guidelines for the diagnosis and management of disseminated intravascular coagulation. British Committee for Standards in Haematology. Br J Haematol. 2009 Apr;145(1):24-33. doi: 10.1111/j.1365-2141.2009.07600.x. Epub 2009 Feb 12. PMID: 19222477.
25. Li T, Lu H, Zhang W. Clinical observation and management of COVID-19 patients. Emerg Microbes Infect. 2020 Dec;9(1):687-690. doi: 10.1080/22221751.2020.1741327. PMID: 32208840; PMCID: PMC7103696.
26. Tahir Huyut M, Huyut Z, İlkbahar F, Mertoğlu C. What is the impact and efficacy of routine immunological, biochemical and hematological biomarkers as predictors of COVID-19 mortality? Int Immunopharmacol. 2022 Apr;105:108542. doi: 10.1016/j.intimp.2022.108542. Epub 2022 Jan 17. Erratum in: Int Immunopharmacol. 2023 Oct;123:110821. PMID: 35063753; PMCID: PMC8761578
27. Zhao Q, Meng M, Kumar R, Wu Y, Huang J, Deng Y, Weng Z, Yang L. Lymphopenia is associated with severe coronavirus disease 2019 (COVID-19) infections: A systemic review and meta-analysis. Int J Infect Dis. 2020 Jul;96:131-135. doi: 10.1016/j.ijid.2020.04.086. Epub 2020 May 4. PMID: 32376308; PMCID: PMC7196544.
28. Tan L, Wang Q, Zhang D, Ding J, Huang Q, Tang YQ, Wang Q, Miao H. Lymphopenia predicts disease severity of COVID-19: a descriptive and predictive study. Signal Transduct Target Ther. 2020 Mar 27;5(1):33. doi: 10.1038/s41392-020-0148-4. Erratum in: Signal Transduct Target Ther. 2020 Apr 29;5(1):61. PMID: 32296069; PMCID: PMC7100419.
29. Bhatraju PK, Ghassemieh BJ, Nichols M, Kim R, Jerome KR, Nalla AK, Greninger AL, Pipavath S, Wurfel MM, Evans L, Kritek PA, West TE, Luks A, Gerbino A, Dale CR, Goldman JD, O'Mahony S, Mikacenic C. Covid-19 in Critically Ill Patients in the Seattle Region - Case Series. N Engl J Med. 2020 May 21;382(21):2012-2022. doi: 10.1056/NEJMoa2004500. Epub 2020 Mar 30. PMID: 32227758; PMCID: PMC7143164.
30. Zhang JJ, Cao YY, Tan G, Dong X, Wang BC, Lin J, Yan YQ, Liu GH, Akdis M, Akdis CA, Gao YD. Clinical, radiological, and laboratory characteristics and risk factors for severity and mortality of 289 hospitalized COVID-19 patients. Allergy. 2021 Feb;76(2):533-550. doi: 10.1111/all.14496. Epub 2020 Aug 24. PMID: 32662525; PMCID: PMC7404752.
31. : https://eody.gov.gr/wp-content/uploads/2022/04/covid_19_algorithmos-mi-nosileuomenon_20220404.pdf

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 18 years old,
2. Hospital treatment for more than 24 hours for SARS-COV -2 infection, confirmed by molecular testing (rRT - PCR) and within one (1) month of the positive test for covid-19 diagnosis.

Exclusion Criteria:

Patients with myelodysplastic syndrome, iron deficiency or low values of B12, folic acid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected by COVID-19
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Survival of patients | 1 month
  Our study will examine the relationship of the red cell index RDW, platelet count PLTs and platelet index MPV/PLT ratio, with the risk of mortality in hospitalized patients with SARS-COV2, at entry, discharge, 1st week , 2nd week, as well as the total duration of hospitalization. There are no other reports on this issue in Greece.

CONTACTS AND LOCATIONS:
Overall Officials: Despoina Georgiadou, MD, Principal Investigator — Sismanogleio Hospital, Sismanogliou 1, Marousi 151 26, Athens, Greece. Amalia Fleming Clinical Unit/ Hematology Department, 25 Martiou, 14, Melissia, 15127, Athens,Greece.
Locations (1):
- Sismanoglio - Amalia Fleming General Hospital/ A.Fleming Clinical Unit, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Anonymized patient data will be provided upon a request to the principal investigator
Supporting Information: Study Protocol, SAP
Time Frame: By 30 June uploaded on ClinicalTrials.org

REFERENCES:
- [Background] Karampitsakos T, Akinosoglou K, Papaioannou O, Panou V, Koromilias A, Bakakos P, Loukides S, Bouros D, Gogos C, Tzouvelekis A. Increased Red Cell Distribution Width Is Associated With Disease Severity in Hospitalized Adults With SARS-CoV-2 Infection: An Observational Multicentric Study. Front Med (Lausanne). 2020 Dec 11;7:616292. doi: 10.3389/fmed.2020.616292. eCollection 2020. PMID 33363191
- [Background] Foy BH, Carlson JCT, Reinertsen E, Padros I Valls R, Pallares Lopez R, Palanques-Tost E, Mow C, Westover MB, Aguirre AD, Higgins JM. Association of Red Blood Cell Distribution Width With Mortality Risk in Hospitalized Adults With SARS-CoV-2 Infection. JAMA Netw Open. 2020 Sep 1;3(9):e2022058. doi: 10.1001/jamanetworkopen.2020.22058. PMID 32965501
- [Background] Atik D, Kaya HB. EVALUATION OF THE RELATIONSHIP OF MPV, RDW AND PVI PARAMETERS WITH DISEASE SEVERITY IN COVID-19 PATIENTS. Acta Clin Croat. 2021 Mar;60(1):103-114. doi: 10.20471/acc.2021.60.01.15. PMID 34588729
- [Background] Azab B, Torbey E, Singh J, Akerman M, Khoueiry G, McGinn JT, Widmann WD, Lafferty J. Mean platelet volume/platelet count ratio as a predictor of long-term mortality after non-ST-elevation myocardial infarction. Platelets. 2011;22(8):557-66. doi: 10.3109/09537104.2011.584086. Epub 2011 Jun 30. PMID 21714700